CLINICAL TRIAL: NCT05180344
Title: Feasibility, Acceptability, and Preliminary Efficacy of a Novel Personalized Mobile Intervention for Suicide
Brief Title: Feasibility, Acceptability, and Preliminary Efficacy of a Novel Personalized Mobile Intervention for Suicide - Open Trial (2)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: American Foundation for Suicide Prevention (AFSP) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1710-001; SRG-1-119-18 (Other Grant/Funding Number: American Foundation for Suicide Prevention])
Record Dates: First submitted 2022-01-03; First posted 2022-01-06 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Suicide; Suicide and Self-harm; Suicide, Attempted; Suicidal Ideation
MeSH Terms: conditions — Suicide; Self-Injurious Behavior; Suicide, Attempted; Suicidal Ideation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile Application to Prevent Suicide (MAPS) (Experimental): Participants receiving MAPS will receive the Safety Planning Intervention (SPI) which will be uploaded into the smartphone app. They will be prompted four times per day to complete a brief ecological momentary assessment "check-in" inquiring about their cognitions, affect, and behavior, including suicidal thoughts and behaviors. Based on these responses, they will be provided with coping strategies from their safety plans and from a database of coping strategies created by study staff. They will also have access to emergency phone numbers, the coping strategies database, and can communicate with their study clinician through a text-like interface in the app. They will receive this intervention for one month.
  Interventions: Behavioral: Mobile Application to Prevent Suicide (MAPS)

INTERVENTIONS:
Behavioral: Mobile Application to Prevent Suicide (MAPS) — Safety Planning Intervention, ecological momentary intervention smartphone app system, and bidirectional communication with study clinician.

SUMMARY:
The primary aim of this grant is to conduct pilot testing on a novel personalized mobile intervention for suicide - Mobile Application to Prevent Suicide (MAPS) - and to establish feasibility, acceptability, safety, and primary outcomes (i.e., suicidal ideation and behavior; re-hospitalization).

ELIGIBILITY:
Inclusion Criteria:

* Suicidal ideation and/or suicidal behavior in the past month verified by the C-SSRS
* Between the ages of 18 and 26
* English proficiency
* Comfortable with smartphone technology
* Deemed by the treatment team to be stable enough to complete study procedures

Exclusion Criteria:

* Current psychotic or manic symptoms severe enough to interfere with study procedures

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Research (Recruitment) | Baseline
  Measured by recruitment rate.
Acceptability of Research (Recruitment) | 1 month
  Measured by dropout rate.
Acceptability of Research Procedures | 1 month
  Feedback on qualitative interview
Patient Satisfaction | 1 month
  Measured using the Client Satisfaction Questionnaire, a self-report measure of satisfaction with treatment. Scores range from 8 to 32, with higher scores representing higher satisfaction.
Acceptability of MAPS Intervention | 1 month
  Feedback on qualitative interview.
Satisfaction with MAPS Intervention | 4 weeks
  Measured by protocol completion rate.
Ecological Momentary Assessment (EMA) Adherence | 4 weeks
  Number of assessments completed out of total.

SECONDARY OUTCOMES:
Suicidal Ideation and Behavior | 1 month
  Will be assessed using the Columbia Suicide Severity Rating Scale, items from the Modified Scale for Suicidal Ideation, and ecological momentary assessment of suicidal ideation and behavior. The Columbia Suicide Severity Rating Scale can provide presence/absence of suicidal ideation and suicidal behavior, as well as a suicidal ideation score ranging from 0 to 5 with higher scores representing more severe ideation, and a suicidal ideation intensity rating from 0-25 with higher scores representing more intense ideation.
Rehospitalization | 1 month
  Will be assessed using the Treatment History Interview and medical records review.

CONTACTS AND LOCATIONS:
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
After all data have been collected and the results of the studies published, de-identified data will be made available to other qualified researchers on request.